CLINICAL TRIAL: NCT03308890
Title: The Effect of Entecavir Consolidation on Post-TDF Treatment Durability
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: China Medical University Hospital (Other); Chang Gung Memorial Hospital (Other); Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, vghtpe user, Professor and Chief of Gastroenterology & Hepatology, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AI463-527
Record Dates: First submitted 2017-10-05; First posted 2017-10-13 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: Arm 1：0.5mg Entecavir QD for 6 months after cessation of TDF. Arm 2：0.5mg Entecavir QD for 12 months after cessation of TDF. Arm 3：No consolidation arm and observation only. Clinical observation for up to 6 months after the end of study follow-up for all arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): 0.5mg Entecavir QD for 6 months after cessation of TDF and clinical observation for up to 6 months after the end of study follow-up.
  Interventions: Drug: 0.5mg Baraclude(entecavir)
- Arm 2 (Active Comparator): 0.5mg Entecavir QD for 12 months after cessation of TDF and clinical observation for up to 6 months after the end of study follow-up.
  Interventions: Drug: 0.5mg Baraclude(entecavir)
- Arm 3 (No Intervention): No consolidation arm and observation only and clinical observation for up to 6 months after the end of study follow-up.

INTERVENTIONS:
Drug: 0.5mg Baraclude(entecavir) — 0.5mg Baraclude (entecavir) QD for 6 months after cessation of TDF.
  Arms: Arm 1
Drug: 0.5mg Baraclude(entecavir) — 0.5mg Baraclude (entecavir) QD for 12 month after cessation of TDF.
  Arms: Arm 2

SUMMARY:
Clinical relapse occurred much earlier and tended to be more severe after cessation of TDF than ETV. The follow-up interval and intensity would be different between ETV and TDF after discontinuation of therapy. Whether switch therapy from TDF to ETV can modify the pattern of relapse is interesting but unclear. Our hypothesis is that entecavir consolidation on post-TDF treatment patients reduce and delay the clinical relapse effectively. Hence in this proof of concept study we would like to evaluate the effect of 6 months and 12 months of entecavir consolidation on post-TDF treatment durability.

DETAILED DESCRIPTION:
Long term nucleoside/nucleotide analogues (NAs) treatment is required in the treatment of chronic hepatitis B (CHB). According to current treatment guidelines from APASL 2015, NAs treatment can be stopped if, after HBsAg loss following either anti-HBs seroconversion or at least 12 months of a post-HBsAg clearance consolidation period or after treatment for at least 2 years with undetectable HBV DNA documented on three separate occasions, 6 months apart. In Taiwan, the National Health Insurance system only reimburse 3 years NAs for CHB patients. Previous study from Jeng et al. suggested that the 1-year rate of clinical relapse (HBV DNA>2,000 IU/mL plus ALT>2X ULN) after cessation of entecavir(ETV) therapy by APASL stopping rule (treatment >2 years, HBV DNA undetectable >1 year) in HBeAg-negative chronic hepatitis B(CHB) patients was 45%, of which 25.6% occurred within 6 months. Recently, another study from Jeng et al showed that 34 HBeAg(-) patients who stopped TDF therapy by APASL stopping rule were followed-up every 1-3 months for >6 months. Of these 34 patients, mean age was 51.8 years, 82.4% were males and 14(41.2%) were cirrhotic. The 1-year cumulative clinical relapse rate was 46%, of which 93.3% occurred within 6 months, and 13.3% developed decompensation. Clinical relapse occurred much earlier and tended to be more severe after cessation of TDF than ETV. The follow-up interval and intensity would be different between ETV and TDF after discontinuation of therapy. Whether switch therapy from TDF to ETV can modify the pattern of relapse is interesting but unclear. Our hypothesis is that entecavir consolidation on post-TDF treatment patients reduce and delay the clinical relapse effectively. Hence in this proof of concept study we would like to evaluate the effect of 6 months and 12 months of entecavir consolidation on post-TDF treatment durability.

ELIGIBILITY:
Inclusion Criteria:

* >20 yrs old.
* No history of Lamivudine or telbivudine resistance.
* HBsAg positive for more than 6 months.
* HBeAg (-).
* HBeAg-negative CHB under TDF treatment for mora than 2 years and fulfilled APASL 2012 guideline's stopping rule: HBeAg (-): undetectable HBV DNA on 3 separate occasions at least 6 months apart.

Exclusion Criteria:

* Lamivudine/telbivudine resistance.
* HBeAg (+).
* HIV, HCV co-infection.
* Under immunosuppressant treatment (including steroid and biologics).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical relapse rate. | Up to 24 months.
  Clinical relapse rate (HBV DNA>2000 IU/ml and ALT> 2x ULN) within 6 months after cessation of TDF or ETV consolidation treatment (up to 6 or 12 months on post-TDF therapy).

SECONDARY OUTCOMES:
Severity of ATL flare | Up to 24 months.
  Severity of ATL flare (ALT>5X and 10X) within 6 months after cessation of TDF or ETV consolidation treatment (up to 6 or 12 months on post-TDF therapy).
Liver decompensation incidence | Up to 24 months.
  Liver decompensation incidence (Total bilirubin > 2mg/dl and/or PT prolongation> 3 sec) within 6 months after cessation of TDF or ETV consolidation treatment (up to 6 or 12 months on post-TDF therapy).
Renal function changes | Up to 24 months.
  Renal function changes based on eGFR (monitor per 3m) within 6 months after cessation of TDF or ETV consolidation treatment (up to 6 or 12 months on post-TDF therapy).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Background] Jeng WJ, Sheen IS, Chen YC, Hsu CW, Chien RN, Chu CM, Liaw YF. Off-therapy durability of response to entecavir therapy in hepatitis B e antigen-negative chronic hepatitis B patients. Hepatology. 2013 Dec;58(6):1888-96. doi: 10.1002/hep.26549. Epub 2013 Oct 17. PMID 23744454
- [Background] Jeng WJ, Chen YC, Sheen IS, Lin CL, Hu TH, Chien RN, Liaw YF. Clinical Relapse After Cessation of Tenofovir Therapy in Hepatitis B e Antigen-Negative Patients. Clin Gastroenterol Hepatol. 2016 Dec;14(12):1813-1820.e1. doi: 10.1016/j.cgh.2016.07.002. Epub 2016 Jul 9. PMID 27404969